CLINICAL TRIAL: NCT06503107
Title: A Multicenter Clinical Study on the Safety and Efficacy of Nanobody-based Biepitope CAR-T Cells Targeting BCMA in the Treatment of Relapsed/Refractory Multiple Myeloma
Brief Title: Nanobody-based Biepitope CAR-T Cells Targeting BCMA in the Treatment of R/RMM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry); Huazhong University of Science and Technology Union Shenzhen Hospital (Unknown); The Seventh Affiliated Hospital of Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, MEI HENG, : Proferssor, Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: biepitope BCMA CAR-T
Record Dates: First submitted 2024-06-17; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
Keywords: CAR-T; BCMA; Relapsed / Refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effective of nanobody-based biepitope BCMA-targeting CAR-T cells (Experimental): The recommended reinfusion dose of biepitope BCMA-targeting CAR-T cells in this trial is: 1 × 10^6/kg, 2 × 10^6/kg CAR-T cells.
  Interventions: Drug: Nanobody-based biepitope BCMA-targeting CAR-T cells

INTERVENTIONS:
Drug: Nanobody-based biepitope BCMA-targeting CAR-T cells — Each patient will receive nanobody-based biepitope BCMA-targeting CAR-T cell by intravenous infusion on day 0.

SUMMARY:
To explore the safety and efficacy of nanobody-based BCMA-targeting biepitope CAR-T cells in the treatment of relapsed/refractory multiple myeloma，this study will be conducted in multiple study centers, with 60 patients openly enrolled to receive CAR-T cell therapy. Patients participating in clinical trials will be tested and evaluated for treatment safety, efficacy, duration of response, and long-term survival.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, prospective, single-arm clinical study with patients with relapsed/refractory multiple myeloma as the test subjects, in order to evaluate the safety and efficacy of nanobody-based biepitope CAR-T cells targeting BCMA in the treatment of R/RMM, and to collect CAR-T PK/PD indicators. The structure of BCMA target CAR-T is designed to identify two different epitopes of BCMA protein with two recognition domains, in order to killig MM cells without secreting more pro-inflammatory factors and avoiding escape caused by the limitations of single BCMA antigen recognition.

ELIGIBILITY:
Inclusion Criteria:

* Patient or his or her legal guardian voluntarily participates in and signs an informed consent form.
* Aged ≥ 18 years and ≤ 75 years.
* Diagnosed as Multiple Myeloma (MM) according to the international standard for multiple myeloma (IMWG 2014).
* Diagnosed as relapsed/refractory disease or primary refractory disease; relapse is defined as disease progression within 60 days of the most recent treatment with three or more lines of therapy with different mechanisms of action; refractory is defined as failure to achieve MR or above efficacy with prior treatment and disease progression with recent treatment, or disease progression within 60 days of treatment.
* Flow cytometry or immunohistochemistry showed positive BCMA expression in myeloma cells.
* Have not been treated with antibody-based drugs within 2 weeks prior to cell therapy.
* ECOG score 0-2 points.
* HGB≥70g/L，PLT≥30×10^9/L.
* Liver, kidney and cardiopulmonary functions meet the following requirements:

  1. Serum creatinine ≤ 1.5× ULN or creatinine clearance (Cockcroft-Gault) >30 ml/min；
  2. Left ventricular ejection fraction (LVEF) ≥50%,
  3. Baseline peripheral oxygen saturation > 90%;
  4. Total bilirubin ≤ 1.5×ULN; ALT and AST ≤2.5×ULN.

Exclusion Criteria:

* Previous diagnosis and treatment of other malignancies within 3 years;
* Presence of one of the following cardiac criteria: atrial fibrillation; Myocardial infarction within the last 12 months; Prolonged QT syndrome or secondary QT prolongation, as judged by the investigator. Echocardiogram LVSF <30% or LVEF <50%; Clinically significant pericardial effusion; Cardiac insufficiency NYHA (New York Heart Association) III or IV (absence of this symptom confirmed by echocardiography within 12 months of treatment);
* Patients with active GVHD;
* Patients with a history of severe pulmonary impairment disease;
* Combined with other malignant tumors in the advanced stage;
* Co-infection with severe or persistent infection that cannot be effectively controlled;
* Combined with severe autoimmune disease or congenital immunodeficiency;
* Active hepatitis (hepatitis B virus deoxyribonucleic acid [HBV-DNA ≥ 500 IU/ml and abnormal liver function] or hepatitis C antibody [HCV-Ab] positive, HCV-RNA above the lower limit of detection of the analytical method and abnormal liver function);
* Human immunodeficiency virus (HIV) infection or syphilis infection;
* Patients with a history of severe allergy to biological products (including antibiotics);
* Patients with central nervous system disorders such as uncontrolled epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, etc;
* Pregnant or Lactating Women; Patients and his or her spouses have a fertility plan within 12 months after CAR-T cell infusion;
* Other conditions considered inappropriate by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2026-10-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | within 3 years after infusion
  Therapy-related adverse events (AE), including severe adverse events (SAE) and laboratory outliers with clinical significance, will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
Overall response rate (ORR) of nanobody-based biepitope CAR-T cells targeting BCMA in R/R MM | within 3 years after infusion
  Disease overall response rate (ORR) will be assessed from CAR-T cell infusion to death or last follow-up (censored).
  The rates of stringent complete response (sCRs), complete response (CR), very good partial response (VGPR), partial response (PR), minimal response (MR) will be assessed from CAR T cell infusion to death or last follow-up (censored). ORR will be assessed from CAR T cell infusion to death or last follow-up.
The rates of complete response (CR) of nanobody-based biepitope CAR-T cells targeting BCMA in R/R MM | within 3 years after infusion
  CR will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Very good partial response (VGPR) of nanobody-based biepitope CAR-T cells targeting BCMA in R/R MM | within 3 years after infusion
  VGPR will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Partial response rate (PR) of nanobody-based biepitope CAR-T cells targeting BCMA in R/R MM | within 3 years after infusion
  PR will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Stable diseases (SD) of nanobody-based biepitope CAR-T cells targeting BCMA in R/R MM | within 3 years after infusion
  SD will be assessed from CAR-T cell infusion to death or last follow-up (censored).

SECONDARY OUTCOMES:
Overall survival (OS) of nanobody-based biepitope CAR-T cells targeting BCMA in Relapsed/Refractory multiple myeloma | within 3 years after infusion
  OS will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Progression-free survival (PFS) of nanobody-based biepitope CAR-T cells targeting BCMA in Relapsed/Refractory multiple myeloma | within 3 years after infusion
  PFS will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Event-free survival (EFS) of nanobody-based biepitope CAR-T cells targeting BCMA in Relapsed/Refractory multiple myeloma | within 3 years after infusion
  EFS will be assessed from CAR-T cell infusion to death or last follow-up (censored).

OTHER OUTCOMES:
In vivo expansion and survival of nanobody-based biepitope CAR-T cells targeting BCMA | within 3 years after infusion
  Quantity of CAR copies in bone marrow, peripheral blood and cerebrospinal fluid will be determined by using flow cytometry and quantitative polymerase chain reaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Cohen AD, Garfall AL, Stadtmauer EA, Melenhorst JJ, Lacey SF, Lancaster E, Vogl DT, Weiss BM, Dengel K, Nelson A, Plesa G, Chen F, Davis MM, Hwang WT, Young RM, Brogdon JL, Isaacs R, Pruteanu-Malinici I, Siegel DL, Levine BL, June CH, Milone MC. B cell maturation antigen-specific CAR T cells are clinically active in multiple myeloma. J Clin Invest. 2019 Mar 21;129(6):2210-2221. doi: 10.1172/JCI126397. PMID 30896447
- [Background] Berdeja JG, Madduri D, Usmani SZ, Jakubowiak A, Agha M, Cohen AD, Stewart AK, Hari P, Htut M, Lesokhin A, Deol A, Munshi NC, O'Donnell E, Avigan D, Singh I, Zudaire E, Yeh TM, Allred AJ, Olyslager Y, Banerjee A, Jackson CC, Goldberg JD, Schecter JM, Deraedt W, Zhuang SH, Infante J, Geng D, Wu X, Carrasco-Alfonso MJ, Akram M, Hossain F, Rizvi S, Fan F, Lin Y, Martin T, Jagannath S. Ciltacabtagene autoleucel, a B-cell maturation antigen-directed chimeric antigen receptor T-cell therapy in patients with relapsed or refractory multiple myeloma (CARTITUDE-1): a phase 1b/2 open-label study. Lancet. 2021 Jul 24;398(10297):314-324. doi: 10.1016/S0140-6736(21)00933-8. Epub 2021 Jun 24. PMID 34175021
- [Result] Lee DW, Kochenderfer JN, Stetler-Stevenson M, Cui YK, Delbrook C, Feldman SA, Fry TJ, Orentas R, Sabatino M, Shah NN, Steinberg SM, Stroncek D, Tschernia N, Yuan C, Zhang H, Zhang L, Rosenberg SA, Wayne AS, Mackall CL. T cells expressing CD19 chimeric antigen receptors for acute lymphoblastic leukaemia in children and young adults: a phase 1 dose-escalation trial. Lancet. 2015 Feb 7;385(9967):517-528. doi: 10.1016/S0140-6736(14)61403-3. Epub 2014 Oct 13. PMID 25319501
- [Result] Ali SA, Shi V, Maric I, Wang M, Stroncek DF, Rose JJ, Brudno JN, Stetler-Stevenson M, Feldman SA, Hansen BG, Fellowes VS, Hakim FT, Gress RE, Kochenderfer JN. T cells expressing an anti-B-cell maturation antigen chimeric antigen receptor cause remissions of multiple myeloma. Blood. 2016 Sep 29;128(13):1688-700. doi: 10.1182/blood-2016-04-711903. Epub 2016 Jul 13. PMID 27412889